CLINICAL TRIAL: NCT02827266
Title: NADIR: Multicentre, Open-Label Trial Evaluating a Simple NeoRecormon Regimen in Anemic Patients With Diabetes and Chronic Kidney Disease (Stage 2 to 5) Who Are Not on Dialysis
Brief Title: A Study of Epoetin Beta (NeoRecormon) in Anemic Participants With Diabetes and Chronic Renal Failure Who Are Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18730
Record Dates: First submitted 2016-04-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin beta (Experimental): Participants will receive epoetin beta over an 8-week correction phase and a 4-week extension or continuation phase, for a total exposure of up to 12 weeks.
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — Participants will receive epoetin beta as a weekly subcutaneous (SC) injection over an 8-week correction phase with 60 international units per kilograms (IU/kg) as starting dose. Baseline weight will be used to determine the dose and adjustments in the dose will be implemented based on the participant's blood hemoglobin levels. Participants with a response to correction treatment will then enter a 4-week extension phase to receive the SC injection every 2 weeks, and those without response will continue at the same weekly dose for a 4-week continuation phase.
  Other Names: NeoRecormon and RO 205-3859

SUMMARY:
This study will evaluate the effect of epoetin beta (NeoRecormon) on correction of anemia and quality of life in participants with diabetes and chronic renal failure and who are not receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* Chronic renal failure (stage 2 to stage 5) defined by Glomerular Filtration Rate (GFR) less than (<) 90 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2)
* Anemia related to chronic kidney disease and requiring treatment with erythropoiesis-stimulating agent (ESA) (2 values of hemoglobin less than or equal to 11 gram per deciliter [g/dL] during the 3 months prior to inclusion), and hemoglobin greater than 8 g/dL

Exclusion Criteria:

* Anemia due to a non-renal cause
* Poorly controlled hypertension
* Treatment with an erythropoiesis stimulating agent (ESA) within 3 months prior to the study
* Planned dialysis in next 3 months or organ transplant
* History of cancer except for basal cell cancer and cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Hemoglobin Greater Than (>) 11 Grams per Deciliter (g/dL) After 8-Week Correction Phase | Week 8

SECONDARY OUTCOMES:
Percentage of Participants With Hemoglobin >11 g/dL After 4-Week Extension Phase | Week 12
Percentage of Participants With Hemoglobin >11 g/dL After 4-Week Continuation Phase | Week 12
Quality of Life of Participants as Assessed From Short Form 36 (SF-36) Scores | Baseline, Week 8, 12
Percentage of Participants With Positive Response to Questionnaire for Practicality and Safety of Self-administration of Study Drug | Week 8, 12
Number of Participants With Local Injection Site Reactions | Up to 12 weeks
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 12 weeks
Number of Participants With Chronic Kidney Disease | Baseline
Response to Treatment at the end of the Correction Phase Among Participants With Different Time Since Diabetes Diagnosis | Week 8
Response to Treatment at the end of the Correction Phase Among Participants With Different Hemoglobin Levels at Baseline | Week 8
Response to Treatment at the end of the Correction Phase Among Participants With Different Hematocrit at Baseline | Week 8
Number of Participants per Category of History of Medical Disorders and Surgical Procedures | Baseline
Number of Participants per Type of Diabetes | Week 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (73):
- France (73):
  - Aix-en-Provence
  - Angers
  - Annonay
  - Arras
  - Aubervilliers
  - Beauvais
  - Besançon
  - Béziers
  - Blois
  - Bois-Bernard
  - Bois-Guillaume
  - Bordeaux
  - Boulogne
  - Bourg-en-Bresse
  - Bourgoin
  - Brivé
  - Cabestany
  - Chamalières
  - Chartres
  - Clermont-Ferrand
  - Colmar
  - Creil
  - Créteil
  - Dijon
  - Évian-les-Bains
  - Évreux
  - Évry
  - Figanières
  - Gap
  - Greize
  - Haguenau
  - Harfleur
  - La Roche-sur-Yon
  - La Tronche
  - Le Havre
  - Le Kremlin-Bicêtre
  - Le Mans
  - Lille
  - Limoges
  - Marseille
  - Martigues
  - Maubeuge
  - Melun
  - Mont-de-Marsan
  - Montpellier
  - Montreuil
  - Muret
  - Nevers
  - Niort
  - Nîmes
  - Orléans
  - Paris
  - Pierre-Bénite
  - Poissy
  - Poitiers
  - Quimper
  - Reims
  - Rouen
  - Saint-Brieuc
  - Saint-Laurent-du-Var
  - Saint-Lô
  - Saint-Maurice
  - Saintes
  - Salouël
  - Sens
  - Thiais
  - Thionville
  - Toulouse
  - Tournan-en-Brie
  - Trappes
  - Valence
  - Valenciennes
  - Vandœuvre-lès-Nancy